CLINICAL TRIAL: NCT07023614
Title: A Global Phase 2b, Randomized, Double-Blinded, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Ninerafaxstat in Patients With Symptomatic Non-Obstructive Hypertrophic Cardiomyopathy - FORTITUDE-HCM
Brief Title: A Trial to Evaluate the Efficacy and Safety of Ninerafaxstat in Patients With Symptomatic Non-obstructive Hypertrophic Cardiomyopathy
Acronym: FORTITUDE-HCM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imbria Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMB101-010
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non-obstructive Hypertrophic Cardiomyopathy
Keywords: nHCM; non-obstructive HCM; non-obstructive hypertrophic cardiomyopathy; HCM; hypertrophic cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ninerafaxstat (Experimental)
  Interventions: Drug: Ninerafaxstat 200mg MR
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ninerafaxstat 200mg MR — Ninerafaxstat 200mg Modified Release tablet administered BID
  Arms: Ninerafaxstat
Drug: Placebo — Matching placebo tablet administered BID
  Arms: Placebo

SUMMARY:
FORTITUDE-HCM is a global, multicenter, double-blind, parallel-group, placebo-controlled Phase 2b study that will assess the efficacy and safety of ninerafaxstat compared to placebo on top of Standard of Care in patients with symptomatic nHCM

ELIGIBILITY:
Select Inclusion Criteria:

* Has a clinical diagnosis of HCM consistent with current American College of Cardiology/American Heart Association and European Society of Cardiology Guideline definitions
* Has had confirmation of nHCM by the echocardiography core laboratory based on screening rest and exercise stress echocardiography
* New York Heart Association (NYHA) functional Class II or III at screening
* Functional limitation as defined by a screening CPET

Select Exclusion Criteria:

* Has a known or suspected infiltrative, genetic, or storage disorder causing cardiac hypertrophy that mimics nHCM
* Has any other condition judged by the investigator to be the primary cause of dyspnea, exercise intolerance, and/or angina
* Has an inability to exercise on a treadmill or bicycle (eg, orthopedic limitations)
* Has any medical condition that precludes upright exercise stress testing

Other protocol-defined inclusion and exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CSS) | Baseline to Week 12
  The Clinical Summary Score is a merging of symptom frequency and symptom burden domains into a total symptom score combined with the physical limitation domain. Scoring ranges from 0 to 100, with higher scores indicating better health status.

SECONDARY OUTCOMES:
Change in ventilatory efficiency (VE/VCO2 slope) during cardiopulmonary exercise testing (CPET) | Baseline to Week 12
Change in the Kansas City Cardiomyopathy Questionnaire Total Symptom Score (KCCQ-TSS) | Baseline to Week 12
  The Total Symptom Score is a merging of symptom frequency and symptom burden domains. Scoring ranges from 0 to 100, with higher scores indicating better health status.
Change in the Kansas City Cardiomyopathy Questionnaire Physical Limitations Score (KCCQ-PLS) | Baseline to Week 12
  The Physical Limitations Score is a single-domain score. Scoring ranges from 0 to 100, with higher scores indicating better health status.
Change in the Kansas City Cardiomyopathy Questionnaire Overall Summary Score (KCCQ-OSS) | Baseline to Week 12
  The Overall Summary Score is a merging of symptom, physical limitations, social limitations, and quality of life domains. Scoring ranges from 0 to 100, with higher scores indicating better health status.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (9):
  - Imbria Investigational Site, La Jolla, California
  - Imbria Investigational Site, San Francisco, California
  - Imbria Investigational Site, Washington D.C., District of Columbia
  - Imbria Investigational Site, Chicago, Illinois
  - Imbria Investigational Site, Boston, Massachusetts
  - Imbria Investigational Site, Burlington, Massachusetts
  - Imbria Investigational Site, St Louis, Missouri
  - Imbria Investigational Site, Houston, Texas
  - Imbria Investigational Site, Charlottesville, Virginia
- France (3):
  - Imbria Investigational Site, Montpellier
  - Imbria Investigational Site, Paris
  - Imbria Investigational Site, Saint-Herblain
- Imbria Investigational Site, Katowice, Poland
- Portugal (2):
  - Imbria Investigational Site, Guimarães
  - Imbria Investigational Site, Lisbon
- Spain (5):
  - Imbria Investigational Site, Barcelona, Barcelona
  - Imbria Investigational Site, A Coruña, Galicia
  - Imbria Investigational Site, Madrid, Madrid
  - Imbria Investigational Site, Vigo, Pontevedra
  - Imbria Investigational Site, Seville, Sevilla
- United Kingdom (2):
  - Imbria Investigational Site, London, England
  - Imbria Investigational Site, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: Undecided